CLINICAL TRIAL: NCT03668561
Title: Evaluation of the Effect of the CALIGALOC Orthosis on Standing and Walking of Hemiparetic Patients With Ankle Varus
Brief Title: the Effect of the CALIGALOC Orthosis on Standing and Walking of Hemiparetic Patients With Ankle Varus
Acronym: CALIGALOC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017_01; 2017-A02098-45 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-08-01; First posted 2018-09-12 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-08

CONDITIONS: Hemiparesis; Varus Deformity of Equine Carpus
Keywords: stroke; hemiplegia
MeSH Terms: conditions — Paresis; Stroke; Hemiplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (CALIGALOC) (Experimental): Wearing of the Caligaloc orthosis
  Interventions: Device: Caligaloc

INTERVENTIONS:
Device: Caligaloc — 15 days of wearing of the Caligaloc orthosis

SUMMARY:
To assess the benefit of an anti-varus ankle foot orthosis (CALIGALOC, Bauerfeind) on gait and balance parameters in hemiparetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Hemiparesis at > 3 months (whatever the etiology)
* varus or equinovarus foot disturbing the stance phase of gait
* Able to walk at least 10m, with or without assistive device

Exclusion Criteria:

* unable to walk 10m
* Botulinum toxin injection less than 3 months before inclusion
* history of neurological or locomotor pathology in addition to the etiology of hemiparesis
* Severe comprehension troubles
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-02-22 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
10-meter walk test (in seconds) | comparison between baseline and 15 days
  Maximum gait velocity, from a standing start

SECONDARY OUTCOMES:
Assessment of gait temporospatial parameters by GaitRite® | comparison between baseline and 15 days
  Specific temporal and spatial parameters of gait will be measured with the GaitRite gait evaluation system: gait cadence, hemiparetic step length, spatial asymmetry, swing and stance times.
Posturographic analysis during static upright stance (center of pressure surface) | comparison between baseline and 15 days
  Assessment of displacements of the center of pressure during quiet upright standing for 30s, using a Zebris platform
Baropodometric analysis during gait | comparison between baseline and 15 days
  Assessment of the paretic footprint during gait, using the Zebris platform
Gait endurance (2-minute walk test) | comparison between baseline and 15 days
  Assessment of maximum gait perimeter during a 2mwt
Assessment of walking function | comparison between baseline and 15 days
  Lower Limb Function assessment scale (LL-FAS, Allart et al. 2015) functional subscores
Tolerability of the wearing of the Caligaloc orthosis assessed by visual analog scale | at 15 days
  visual analog scale (0=major discomfort - 10=excellent comfort)

CONTACTS AND LOCATIONS:
Overall Officials: Etienne Allart, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Swynghedau, CHI, Lille, France